CLINICAL TRIAL: NCT05353556
Title: Effects of Home-based Inspiratory Muscle Training in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Effects of Home-based Inspiratory Muscle Training in Patients With IPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ridvan Aktan, Principal Investigator, PhD, Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RidvanAktan_2022/04-03
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Idiopathic Pulmonary Fibrosis; IPF
Keywords: idiopathic pulmonary fibrosis; inspiratory muscle training; home-based; rehabilitation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: This study was designed as a prospective and experimental study. Participants were randomly divided into two groups; a study group and a control group. The study group will perform inspiratory muscle training at 50% of maximal inspiratory pressure (MIP), and the control group received sham training for 8 weeks.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Patients who perform inspiratory muscle training (IMT) with %50 loading
  Interventions: Device: Inspiratory Muscle Training (IMT)
- Sham Group (Sham Comparator): Patients who perform Sham IMT
  Interventions: Device: Sham IMT

INTERVENTIONS:
Device: Inspiratory Muscle Training (IMT) — The IMT protocol will consist of home-based high-intensity daily training - two cycles of 30 breaths with a 1-min rest between sets, twice a day for 8 weeks using an IMT Threshold device (Threshold IMT Philips® Respironics, Inc). The intensity of the training will be set to 50% of each patient's maximal inspiratory pressure measured every week and was adjusted weekly based on the modified Borg scale from 4 to 6 regarding respiratory effort performed during the session.
  Arms: Study Group
Device: Sham IMT — The IMT protocol will consist of home-based daily training - two cycles of 30 breaths with a 1-min rest between sets, twice a day for 8 weeks using an IMT Threshold device (Threshold IMT Philips® Respironics, Inc). The intensity of the training will be set to the lowest intensity of the IMT Threshold device.
  Arms: Sham Group

SUMMARY:
The aim of this study is to investigate the effects of the home-based inspiratory muscle training program on lung functions, dyspnea, inspiratory muscle strength, functional capacity and quality of life in patients with idiopathic pulmonary fibrosis. Patients are evaluated before the inspiratory muscle training and after 8 weeks of training.

DETAILED DESCRIPTION:
The IMT protocol consisted of home-based high-intensity daily training - two cycles of 30 breaths with a 1-min rest between sets, twice a day for 8 weeks using an IMT Threshold device (Threshold IMT Philips® Respironics, Inc). The intensity of the training was set to 50% of each patient's maximal inspiratory pressure measured every week and was adjusted weekly based on the modified Borg scale from 4 to 6 regarding respiratory effort performed during the session. Patients are evaluated before the inspiratory muscle training and after 8 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosing Idiopathic Pulmonary Fibrosis by a pulmonologist;
* Aged between 40 and 75 years;
* Volunteering to research;
* Stable clinical condition (same medication routine and/or no acute exacerbation in the last for the last 4 weeks).

Exclusion Criteria:

* Inability of the participant to understand or perform the procedures proposed during the evaluations or training program.
* Participating in any pulmonary rehabilitation programs;
* A previous pneumonectomy or lobectomy operation;
* Pneumonia in the last 4 weeks;
* Any pulmonary infection during the study;
* Requirement for supplemental oxygen therapy while resting.
* Having Covid-19 disease (during the study or in the past)
* Orthopaedic or neurological conditions affecting the ability to independent walking

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Change in inspiratory muscle strength | 8 weeks
  MIP

SECONDARY OUTCOMES:
Change in percentages of forced expiratory volume in one second | 8 weeks
  Lung function tests: Percentages of forced expiratory volume in one second (FEV1).
Change in percentages of forced vital capacity | 8 weeks
  Lung function tests: Percentages of forced vital capacity (FVC).
Change in diffusing capacity of the lung for carbon monoxide | 8 weeks
  Lung function tests: Diffusing capacity of the lung for carbon monoxide (DLCO).
Change in Dyspnea | 8 weeks
  The modified Medical Research Council (mMRC) Dyspnea Scale was used to evaluate the severity of dyspnea. Commonly used in the assessment of dyspnea in COPD, mMRC has a five-level scoring system ranging from 0 to 4. A high score indicates an increased sense of dyspnea.
Change in Functional capacity | 8 weeks
  Maximal distance in 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Rıdvan Aktan, PhD, Principal Investigator — Izmir University of Economics
Locations (1):
- Dokuz Eylul University, Izmir, Balcova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Selman M, Thannickal VJ, Pardo A, Zisman DA, Martinez FJ, Lynch JP 3rd. Idiopathic pulmonary fibrosis: pathogenesis and therapeutic approaches. Drugs. 2004;64(4):405-30. doi: 10.2165/00003495-200464040-00005. PMID 14969575
- [Background] Jastrzebski D, Kozielski J, Zebrowska A. [Pulmonary rehabilitation in patients with idiopathic pulmonary fibrosis with inspiratory muscle training]. Pneumonol Alergol Pol. 2008;76(3):131-41. Polish. PMID 18843927
- [Background] Kagaya H, Takahashi H, Sugawara K, Kasai C, Kiyokawa N, Shioya T. Effective home-based pulmonary rehabilitation in patients with restrictive lung diseases. Tohoku J Exp Med. 2009 Jul;218(3):215-9. doi: 10.1620/tjem.218.215. PMID 19561392
- [Background] Tzanakis N, Samiou M, Lambiri I, Antoniou K, Siafakas N, Bouros D. Evaluation of health-related quality-of-life and dyspnea scales in patients with idiopathic pulmonary fibrosis. Correlation with pulmonary function tests. Eur J Intern Med. 2005 Apr;16(2):105-112. doi: 10.1016/j.ejim.2004.09.013. PMID 15833676
- [Background] Peng S, Li Z, Kang J, Hou X. Cross-sectional and longitudinal construct validity of the Saint George's Respiratory Questionnaire in patients with IPF. Respirology. 2008 Nov;13(6):871-9. doi: 10.1111/j.1440-1843.2008.01359.x. PMID 18811886